CLINICAL TRIAL: NCT06275711
Title: The Effect of Therapeutic Communication Program on the Psychological State of Children Affected by the Kahramanmaras Earthquake in Türkiye
Brief Title: The Effect of Therapeutic Communication Program on the Psychological State of Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Gizem Çakır, Research Assistant, Gazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 223K003
Record Dates: First submitted 2024-02-05; First posted 2024-02-23 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Psychological
Keywords: children; earthquake; anxiety; affection; psychological resilience
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Pre-test post-test quasi-experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeutic communication (Experimental): Therapeutic communication methods were applied. Pre-test and post-test measurements were made
  Interventions: Behavioral: Therapeutic communication methods

INTERVENTIONS:
Behavioral: Therapeutic communication methods — Drawing pictures, story completion, breathing and relaxation exercises

SUMMARY:
Earthquake is a disaster that causes physical, psychological, social, economic and cultural losses for individuals and affects/interrupts all age groups and normal life. Children are a group that is more affected by the earthquake than other members of the society and are exposed to its long-term effects. Children who have experienced earthquakes and continue to stay in the earthquake zone experience physical, economic, and social problems. In addition, the emotional and psychological development of these children is negatively affected.

Due to the earthquake that occurred on 6 February 2023 affecting 11 provinces in our country, the needs in the field vary. After the acute period (first 1 month), children need psychological support. Problems that cannot be solved in the early period may cause health and behavioural problems in children in later ages and adulthood. In this context, approaching children with appropriate therapeutic communication methods positively affects their psychological well-being and directly affected physical resilience by enabling them to express their emotions.

The aim of the study was to evaluate the effect of therapeutic communication programme on state and trait anxiety levels, psychological resilience, mental health and well-being of children aged 8-12 years affected by the earthquake.

Hypotheses H1. After the therapeutic communication programme, children's State Anxiety Scale scores decrease.

H2. After the therapeutic communication programme, children's Continuance Anxiety Scale scores decrease.

H3. After the therapeutic communication programme, children's Me and My Emotions Scale scores decrease.

H4. After the therapeutic communication programme, children's scores on the Child and Adolescent Psychological Resilience Scale increase.

DETAILED DESCRIPTION:
Sample of the Research However, since children affected by the earthquake need psychological support, all children who are willing to participate in the programme will be included in order to provide the highest benefit. People who meet the research criteria and volunteer to participate in the research will be selected. In order to determine the power of the research, post-hoc power analysis will be performed using G*power 3.1 programme.

Data Collection Tools Child Data Collection Form, Child State-Trait Anxiety Inventory, Me and My Emotions Scale in Children and Adolescents, Child and Adolescent Psychological Resilience Scale will be used to collect the data.

Data Collection The study will be started after the approval of the ethics commission and permission from the organisation. At the beginning of the study, an introductory meeting will be held with the children and families in order to gain a sense of trust in children and information about the programme will be given. After obtaining consent from the children and their families who agreed to participate in the study, the child data collection form will be filled in by the researchers. Child State-Trait Anxiety Scale, I and My Emotions in Children and Adolescents Scale, Child and Adolescent Psychological Resilience Scale pre-tests will be completed by children. While the children are filling out the forms, the researchers will provide support in reading, explaining the incomprehensible statement and marking if requested. Researchers will not give any guidance to children while providing support. Therapeutic Communication Programme will be started with the children included in the study. After the programme is completed, the final tests of the scales completed by the children will be applied.

Implementation of Therapeutic Communication Programme Children and parents will be invited to the container. Children and parents will be informed about the programme. After obtaining verbal consent from the children who want to participate and written consent from their parents, pre-test forms will be applied and physical evaluations will be made. In addition, a one-session training will be organised for the parents. The next day, the 1-week "Therapeutic Communication Programme", which includes 6 modules, will start to be applied to the children. Each module content is planned to last approximately 1 hour. One module will be applied every day. On the 6th day, after the applications are completed, the post-test application of the scales will be carried out.

Ethics of the Research In order to decide on the ethical appropriateness of the research, approval will be obtained by applying to Gazi University Ethics Commission. Then, written permission will be obtained from the relevant institutions. Before the data collection process, the researchers will inform the individuals who agree to participate in the research about the research, and after explaining the purpose of the research, verbal consent will be obtained from the children and written consent will be obtained from the parents of the children. The research will be conducted in accordance with the principles of the Declaration of Helsinki. Physical assessment (vital signs, posture, assessment of respiration, assessment of bowel movements, assessment of musculoskeletal system, questioning of current disease status, oral examination, skin assessment, cognitive status, etc.) and anthropometric measurements (height and body weight) will be performed in a separate room in the service container. No one other than the child and his/her parent will be allowed in the room.

Data Evaluation Statistical analyses will be performed in IBM SPSS for Windows Version 21.0 package programme. Numerical variables that fit the normal distribution will be analysed by independent groups t-test and one-way analysis of variance (ANOVA). Mann-Whitney U and Kruskal-Wallis tests will be used for comparisons of non-normally distributed numerical measurements. Intergroup comparisons of categorical variables will be analysed by Chi-Square tests. Post-Hoc tests will be used to determine the groups that create the difference in comparisons with significant differences. For all hypothesis tests, the statistical significance level will be set as ≤ 0,05.

ELIGIBILITY:
Inclusion Criteria:

* He is willing to participate in the programme,
* Children aged 8-12 years (verbal consent will be obtained from children and written consent will be obtained from their parents).

Exclusion Criteria:

* Children with psychological diagnoses (since exclusion from the group is not ethically appropriate, these children will be allowed to participate in the trainings, but the data obtained will not be included in the sample group).

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
State Anxiety Scale on Children | before the study is started (day 1) / after the study is completed (day 7)
  The score to be obtained from the trait anxiety subsection of the inventory varies between 20-60. The higher the score obtained from the inventory, the higher the level of anxiety.
Trait Anxiety Scale on Children | before the study is started (day 1) / after the study is completed (day 7)
  The score to be obtained from the trait anxiety subsection of the inventory varies between 20-60. The higher the score obtained from the inventory, the higher the level of anxiety.
Me and My Feelings Scale on Children | before the study is started (day 1) / after the study is completed (day 7)
  The score range for emotional difficulties and behavioural difficulties is 0-20 and 0-12, respectively.
Child and Youth Resilience Measure | before the study is started (day 1) / after the study is completed (day 7)
  High scores obtained from the scale indicate a high level of psychological resilience. There is no cut-off value.

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Cakir, PhD(c), Principal Investigator — Gazi University Nursing Faculty; Rukiye Celik, PhD(c), Principal Investigator — Gazi University Nursing Faculty; Naime Altay, PhD, Principal Investigator — Gazi University
Locations (1):
- K-1 Container City, Adıyaman, Altınsehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanc J, Eugene D, Louis EF, Cadichon JM, Joseph J, Pierre A, Laine R, Alexandre M, Huang KY. Mental Health Among Children Older than 10 Years Exposed to the Haiti 2010 Earthquake: a Critical Review. Curr Psychiatry Rep. 2020 Sep 2;22(11):57. doi: 10.1007/s11920-020-01178-9. PMID 32876808
- [Background] Sever MS, Sever L, Vanholder R. Disasters, children and the kidneys. Pediatr Nephrol. 2020 Aug;35(8):1381-1393. doi: 10.1007/s00467-019-04310-x. Epub 2019 Aug 17. PMID 31422466
- See also: Children's earthquake preparedness and risk perception: A comparative study of two cities in Turkey, using a modified PRISM approach — https://doi.org/10.1016/j.ijdrr.2020.101666
- See also: Impact evaluation of a school-based disaster education program in a city affected by the 2011 great East Japan earthquake and tsunami disaster — https://doi.org/10.1016/j.ijdrr.2020.101632